CLINICAL TRIAL: NCT00789828
Title: A Randomized, Double-blind, Placebo-controlled Study of Everolimus in the Treatment of Patients With Subependymal Giant Cell Astrocytomas (SEGA) Associated With Tuberous Sclerosis Complex (TSC)
Brief Title: Efficacy and Safety of Everolimus (RAD001) in Patients of All Ages With Subependymal Giant Cell Astrocytoma Associated With Tuberous Sclerosis Complex (TSC)(EXIST-1)
Acronym: EXIST-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001M2301; 2007-006997-27 (EudraCT Number)
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Tuberous Sclerosis; Subependymal Giant Cell Astrocytoma
Keywords: SEGA; Tuberous Sclerosis; Subependymal Giant Cell Astrocytoma; mTOR; RAD001; Mamalian Target Rapamycin; Everolimus; TSC
MeSH Terms: conditions — Tuberous Sclerosis; Astrocytoma | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Everolimus (Experimental): Everolimus was administered orally at a starting dose of 4.5mg/m^2 daily and subsequently titrated to attain whole blood trough concentration of 5 to 15 ng/mL. Dose adjustments were permitted based on safety and whole blood trough concentrations.
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): Matching Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus was formulated as tablets of 1.0-mg strength and was blisterpacked under aluminum foil in units of 10 tablets.
  Other Names: RAD001
  Arms: Everolimus
Drug: Placebo — Placebo was provided as a matching tablet and was blisterpacked under aluminum foil in units of 10.
  Arms: Placebo

SUMMARY:
This study evaluated the efficacy and safety of Everolimus in treating patients with Subependymal Giant Cell Astrocytomas associated with Tuberous Sclerosis Complex.

ELIGIBILITY:
Inclusion Criteria:

* All Ages
* Definite diagnosis of Tuberous Sclerosis according to the modified Gomez criteria
* At least one Subependymal Giant Cell Astrocytoma of at least 1 cm in diameter
* Evidence of SEGA worsening as compared to prior MRI scans
* Females of child bearing potential must use birth control
* Written informed consent

Exclusion Criteria:

* SEGA related surgery is likely to be required in the opinion of the investigator
* Recent heart attack, cardiac related chest pain or stroke
* Severely impaired lung function
* Severe liver dysfunction
* Severe kidney dysfunction
* Pregnancy or breast feeding
* Current infection
* History of organ transplant
* Surgery within two months prior to study enrollment
* Prior therapy with a medication in the same class as Everolimus
* Uncontrolled high cholesterol
* Uncontrolled diabetes
* HIV
* Patients with metal implants thus prohibiting MRI evaluations

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Tuberous Sclerosis Center, Phoenix, Arizona
  - University of California at Los Angeles, Los Angeles, California
  - Children's Hospital Oakland Hematology/Oncology Dept, Oakland, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of CHicago Comer Children's Hospital, Chicago, Illinois
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Children's Hospital Boston SC-1, Boston, Massachusetts
  - Minnesota Epilepsy Group - PA, Saint Paul, Minnesota
  - Cincinnati Children's Hospital Medical Center Cincinnati Children's Hosp, Cincinnati, Ohio
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Children's Regional Outpatients Center SC, Fairfax, Virginia
- Novartis Investigative Site, Randwick, New South Wales, Australia
- Novartis Investigative Site, Brussels, Belgium
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma
- Novartis Investigative Site, Utrecht, Netherlands, Netherlands
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Bristol, United Kingdom

REFERENCES:
- [Derived] Bissler JJ, Budde K, Sauter M, Franz DN, Zonnenberg BA, Frost MD, Belousova E, Berkowitz N, Ridolfi A, Christopher Kingswood J. Effect of everolimus on renal function in patients with tuberous sclerosis complex: evidence from EXIST-1 and EXIST-2. Nephrol Dial Transplant. 2019 Jun 1;34(6):1000-1008. doi: 10.1093/ndt/gfy132. PMID 30053159
- [Derived] Sparagana S, Franz DN, Krueger DA, Bissler JJ, Berkowitz N, Burock K, Kingswood JC. Pooled analysis of menstrual irregularities from three major clinical studies evaluating everolimus for the treatment of tuberous sclerosis complex. PLoS One. 2017 Oct 12;12(10):e0186235. doi: 10.1371/journal.pone.0186235. eCollection 2017. PMID 29023494
- [Derived] Franz DN, Belousova E, Sparagana S, Bebin EM, Frost MD, Kuperman R, Witt O, Kohrman MH, Flamini JR, Wu JY, Curatolo P, de Vries PJ, Berkowitz N, Niolat J, Jozwiak S. Long-Term Use of Everolimus in Patients with Tuberous Sclerosis Complex: Final Results from the EXIST-1 Study. PLoS One. 2016 Jun 28;11(6):e0158476. doi: 10.1371/journal.pone.0158476. eCollection 2016. PMID 27351628
- [Derived] Jozwiak S, Kotulska K, Berkowitz N, Brechenmacher T, Franz DN. Safety of Everolimus in Patients Younger than 3 Years of Age: Results from EXIST-1, a Randomized, Controlled Clinical Trial. J Pediatr. 2016 May;172:151-155.e1. doi: 10.1016/j.jpeds.2016.01.027. Epub 2016 Feb 6. PMID 26858193
- [Derived] Goyer I, Dahdah N, Major P. Use of mTOR inhibitor everolimus in three neonates for treatment of tumors associated with tuberous sclerosis complex. Pediatr Neurol. 2015 Apr;52(4):450-3. doi: 10.1016/j.pediatrneurol.2015.01.004. Epub 2015 Jan 14. PMID 25682485
- [Derived] Franz DN, Belousova E, Sparagana S, Bebin EM, Frost M, Kuperman R, Witt O, Kohrman MH, Flamini JR, Wu JY, Curatolo P, de Vries PJ, Berkowitz N, Anak O, Niolat J, Jozwiak S. Everolimus for subependymal giant cell astrocytoma in patients with tuberous sclerosis complex: 2-year open-label extension of the randomised EXIST-1 study. Lancet Oncol. 2014 Dec;15(13):1513-1520. doi: 10.1016/S1470-2045(14)70489-9. Epub 2014 Nov 10. PMID 25456370
- [Derived] Kingswood JC, Jozwiak S, Belousova ED, Frost MD, Kuperman RA, Bebin EM, Korf BR, Flamini JR, Kohrman MH, Sparagana SP, Wu JY, Brechenmacher T, Stein K, Berkowitz N, Bissler JJ, Franz DN. The effect of everolimus on renal angiomyolipoma in patients with tuberous sclerosis complex being treated for subependymal giant cell astrocytoma: subgroup results from the randomized, placebo-controlled, Phase 3 trial EXIST-1. Nephrol Dial Transplant. 2014 Jun;29(6):1203-10. doi: 10.1093/ndt/gfu013. Epub 2014 Apr 11. PMID 24729041
- [Derived] Kotulska K, Borkowska J, Jozwiak S. Possible prevention of tuberous sclerosis complex lesions. Pediatrics. 2013 Jul;132(1):e239-42. doi: 10.1542/peds.2012-3607. Epub 2013 Jun 3. PMID 23733802
- [Derived] Franz DN, Belousova E, Sparagana S, Bebin EM, Frost M, Kuperman R, Witt O, Kohrman MH, Flamini JR, Wu JY, Curatolo P, de Vries PJ, Whittemore VH, Thiele EA, Ford JP, Shah G, Cauwel H, Lebwohl D, Sahmoud T, Jozwiak S. Efficacy and safety of everolimus for subependymal giant cell astrocytomas associated with tuberous sclerosis complex (EXIST-1): a multicentre, randomised, placebo-controlled phase 3 trial. Lancet. 2013 Jan 12;381(9861):125-32. doi: 10.1016/S0140-6736(12)61134-9. Epub 2012 Nov 14. PMID 23158522
- See also: Visit EXIST-1 NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/portals/EXISTClinicalTrials/page.do

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 centers in 10 countries.
Pre-assignment Details: A total of 117 participants were enrolled and randomized into the core period. Only 111 participants completing the core period, continued in the open-label extension period of the study.
Groups:
- Everolimus: Participants received oral dose of everolimus 4.5 milligram/square meter (mg/m^2) daily as an initial starting dose to attain the whole blood trough concentrations in range of 5-15 nanogram/millilitre (ng/mL). Dose adjustments were permitted based on safety and whole blood trough concentrations.
- Placebo: Participants received oral dose of placebo matching to everolimus daily.
Period: Core Period (48 Weeks)
Arm/Group | Everolimus | Placebo
Started | 78 | 39
Completed | 78 | 33
Not Completed | 0 | 6
Not completed — Administrative problems | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Period: Open-label Extension Period (4 Years)
Arm/Group | Everolimus | Placebo
Started | 111 (Of 117 participants only 111 completed the core period and continued in the extension period) | 0 (No participant received placebo.)
Completed | 82 | 0
Not Completed | 29 | 0
Not completed — Adverse Event | 10 | 0
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Administrative problems | 7 | 0
Not completed — Death | 1 | 0
Not completed — Disease progression | 1 | 0
Not completed — New treatment for indication under study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Everolimus (Core Period): Participants received oral dose of everolimus 4.5 mg/m^2 daily as an initial starting dose to attain the whole blood trough concentrations in range of 5-15 ng/mL. Dose adjustments were permitted based on safety and whole blood trough concentrations.
- Placebo (Core Period): Participants received oral dose of placebo matching to everolimus daily.
- Total: Total of all reporting groups
Arm/Group | Everolimus (Core Period) | Placebo (Core Period) | Total
Number analyzed (Participants) | 78 | 39 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (5.9) | 10.3 (7.3) | 10.2 (6.4)
Age, Customized [Number; unit: Participants]
  <3 years | 13 | 7 | 20
  3-18 years | 55 | 26 | 81
  ≥18 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 50
  Male | 49 | 18 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Subependymal Giant Cell Astrocytomas (SEGA) Response
Description: Participants were assessed for SEGA response, defined as 50% reduction from baseline in SEGA volume (where SEGA volume was the sum of the volumes of all target SEGA lesions identified at baseline, and confirmed with a second scan performed approximately 12 weeks later), no unequivocal worsening of non-target SEGA lesions, no new SEGA lesions (≥ 1 cm in longest diameter), and no new or worsening hydrocephalus. Multi-phase brain MRI was utilized to identify SEGA lesions. SEGA response rate was defined as the percentage of participants whose best overall status was SEGA response as determined by Independent Central Radiology Review. The Kaplan-Meier estimate was used for determining time to SEGA response.
Time Frame: End of core period (Week 48), and end of extension period (up to 4 years)
Population: The primary analysis was performed in Full Analysis Set (FAS) population, defined as all randomized participants involved in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Everolimus (Extension Period): Participants received oral dose of everolimus 4.5 mg/m^2 daily as an initial starting dose to attain blood trough concentrations in range of 5-15 ng/mL.
Arm/Group | Everolimus (Core Period) | Placebo (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 78 | 39 | 111
Percentage of participants | 34.6 [24.2 to 46.2] | 0.0 [0.0 to 9.0] | 57.7 [47.9 to 67]

2. Secondary Outcome: Change From Baseline in Frequency of Total Seizure Events Per 24 Hours at Week 24 in Both Core and Extension Period
Description: Seizure frequency per 24 hours was defined as the number of seizures in the electroencephalography (EEG) divided by the number of hours in the EEG, multiplied by 24. Seizure frequency was evaluated using a 24-hour video-EEG. Seizure frequency was listed as missing if the actual EEG recording duration was < 18 hours.
Time Frame: Baseline (Core period) to Week 24 (Core period), Baseline (Extension period, Week 24 post-core baseline) to Week 24 (Extension period, Week 48 post-core baseline)
Population: The analysis was performed in the FAS population. Missing values were imputed using last observation carried forward approach for core period while raw count for extension period.
Measure: Mean (Standard Deviation); unit: Seizure frequency
Arm/Group | Everolimus (Core Period) | Placebo (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 78 | 39 | 34
Seizure frequency | -1.24 (6.12) | -0.24 (5.7) | -6.07 (9.719)

3. Secondary Outcome: Time to SEGA Progression
Description: Time to SEGA progression was defined as time between randomisation to time to first SEGA progression. SEGA progression was defined as either one or more of the following criteria: 1. increase from nadir of ≥ 25% in SEGA volume to a value greater than baseline SEGA volume (where SEGA volume is the sum of the volumes of all target SEGA lesions identified at baseline, and nadir is the lowest SEGA volume obtained for the participant previously in the trial), 2. unequivocal worsening of non-target SEGA lesions, 3. appearance of new SEGA lesion ≥ 1.0 cm in longest diameter, 4. new or worsening hydrocephalus. The median TTSP based on central radiology review was not reached in any treatment arms; Only 6 events of SEGA progressions were observed in the placebo group of core period.
Time Frame: Baseline up to week 48 (end of core period), and end of extension period (up to 4 years)
Population: The analysis was performed in the FAS population. Here "Number of participants analysed" signifies the participants assessed for time to SEGA progression during the study for each arm, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus (Core Period) | Placebo (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 78 | 39 | 111
months | NA [NA to NA] — Median was not reached as no participant experienced disease progression during core period. | NA [NA to NA] — Median was not reached as only 6 participants experienced disease progression during core period. | NA [NA to NA] — Median was not reached as no participant experienced disease progression during extension period.

4. Secondary Outcome: Time to SEGA Response
Description: Participants were assessed for time to SEGA response, defined as 50% reduction from baseline in SEGA volume (where SEGA volume was the sum of the volumes of all target SEGA lesions identified at baseline, and confirmed with a second scan performed approximately 12 weeks later), no unequivocal worsening of non-target SEGA lesions, no new SEGA lesions (≥ 1 cm in longest diameter), and no new or worsening hydrocephalus. Multi-phase brain MRI was utilised to identify SEGA lesions. SEGA response rate was defined as the percentage of participants whose best overall status was SEGA response as determined by Independent Central Radiology Review. The Kaplan-Meier estimate was used for determining time to SEGA response.
Time Frame: Baseline up to week 48 (end of core period), and end of extension period (up to 4 years)
Population: The analysis was performed in the FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 27 | 64
months | 2.99 [2.79 to 5.36] | 5.32 [3.02 to 5.59]

5. Secondary Outcome: Duration of SEGA Response
Description: Duration of SEGA response was defined as time from the date of the first documented SEGA response until the date of the first documented SEGA progression. Duration of SEGA response was evaluated only for participants who achieved a SEGA response. The time to SEGA progression was censored if SEGA progression was not observed before the first to occur out of (i) analysis cut-off date (ii) the date when systemic anti-SEGA medication is started, (iii) the date of a SEGA-related surgery or (iv) the date of death. Since, no case of SEGA progression was observed in core study which resulted in censored duration of SEGA response. Only 5 SEGA responders experienced a SEGA progression in extension period.
Time Frame: Baseline up to week 48 (end of core period), and end of extension period (up to 4 years)
Population: The analysis was performed in the FAS population. Here, "Number of participants analysed" signifies the participants assessed for SEGA progression during the study for each arm, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 27 | 64
months | NA [NA to NA] — Median was not achieved as no case of SEGA progression was observed. | NA [NA to NA] — Median was not achieved as only 5 events of SEGA progression were observed.

6. Secondary Outcome: Time to SEGA Worsening
Description: Time to SEGA worsening was defined as the time from the start of everolimus to date of the first SEGA worsening. SEGA worsening was defined as either; increase from nadir of ≥ 25% in SEGA volume or unequivocal worsening of non-target SEGA lesions, or appearance of new SEGA lesion ≥ 1.0 cm in longest diameter, or new or worsening hydrocephalus. The median value was not reached in either treatment arm of core period as SEGA worsening was observed in less participants (everolimus - 7 and placebo - 8).
Time Frame: Baseline up to week 48 (end of core period), and end of extension period (up to 4 years)
Population: The analysis was performed in the FAS population. Here, "Number of participants analysed" signifies the participants assessed for time to SEGA worsening during the study for each arm, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus (Core Period) | Placebo (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 78 | 39 | 111
months | NA [NA to NA] — Median was not achieved as only 7 events of SEGA progression were observed. | NA [NA to NA] — Median was not achieved as only 8 events of SEGA progression were observed. | 55.72 [55.72 to NA] — Median upper value was not available as only single of SEGA progression were observed.

7. Secondary Outcome: Percentage of Participants With Skin Lesions Assessed Using Physician's Global Assessement Overall Score
Description: Skin lesions included hypomelanotic macules, the shagreen patch, periungual or subungual fibromas, facial angiofibromas and/or forehead plaques. Response was evaluated using the Physician's Global Assessment of Clinical Condition (PGA) on a 7-point scale: Grade 0 = complete clinical response, indicated absence of disease, Grade 1, 2, and 3 = partial response, indicated improvements of ≥ 50% but < 100%, Grade 4, 5 = stable disease, indicated some or no improvements of 25% - < 50% and 6 = progressive disease, indicated worse than at baseline evaluation by > 25%. Response rate was determined for participants with ≥ 1 skin lesion at baseline, defined as the percentage of participants with overall status as complete clinical response or partial response.
Time Frame: End of core period (Week 48), and end of extension period (up to 4 years)
Population: The analysis was performed in the FAS population. Here, "Number of participants analysed" signifies the participants assessed for skin lesion response during the study for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus (Core Period) | Placebo (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 72 | 38 | 105
Percentage of participants | 41.7 [30.2 to 53.9] | 10.5 [2.9 to 24.8] | 58.1 [48.1 to 67.7]

8. Secondary Outcome: Duration of Skin Lesion Response in Everolimus Treated Participants
Description: Duration of skin lesion response was defined as the time from the first skin lesion response until the first skin lesion progression, defined as worsening of lesion by > 25% or more from baseline.
Time Frame: Baseline up to week 48 (end of core period), and end of extension period (up to 4 years)
Population: The analysis was performed in the FAS population. Here, "Number of participants analysed" signifies everolimus treated responders with best overall skin lesion response during the core and extension period, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 30 | 61
months | NA [NA to NA] — Median was not achieved as no case of skin lesion was observed. | NA [NA to NA] — Median was not achieved as no case of skin lesion was observed.

9. Secondary Outcome: Everolimus Blood Concentration (C2h) at 2 Hours Post Dose
Description: The participants were assessed for everolimus blood concentration at 2 hours time point after dose administration on the same day, if the participant did not vomit between previous dose and blood sample collection. Tandem liquid chromatography-mass spectrometry method was used for evaluation. C2h values were categorized as < 20 ng/mL, 20-50 ng/mL, and > 50 ng/mL, concentrations below the lower limit of quantification were entered as 0 ng/mL.
Time Frame: 2 hours post dose on Week 6, Week 24, Week 48, Week 96, Week 144, and Week 240
Population: The analysis was performed in the Safety Set population (Only evaluable PK Samples), defined as participants who received at least one dose of the double-blind study drug, with a valid post baseline assessment. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 78 | 111
ng/mL
  Week 6 (n= 37, 47) | 27.52 (15.24) | 27.74 (16.202)
  Week 24 (n= 11, 13) | 38.7 (15.76) | 39.25 (14.662)
  Week 48 (n= 1, 3) | 23.2 (NA) — Only one participant was evaluable, so value was not available. | 49.73 (28.884)
  Week 96 (n= 0, 6) | NA (NA) — No participant was evaluable, so value was not available. | 31.63 (21.902)
  Week 144 (n= 0, 6) | NA (NA) — No participant was evaluable, so value was not available. | 26.33 (11.908)
  Week 240 (n= 0, 0) | NA (NA) — No participant was evaluable, so value was not available. | NA (NA) — No participant was evaluable, so value was not available.

10. Secondary Outcome: Everolimus Trough Concentrations (Cmin) at 24 Hours After Last Dose
Description: The participants were assessed for everolimus trough concentration (Cmin) at 24 hours time point after previous dose administration, at a steady state following 5 days of consistent dosing, if the participant did not vomit within 4 hours of previous dose. Tandem liquid chromatography-mass spectrometry method was used for evaluation. Cmin values were categorized as <5 ng/mL, 5-10 ng/mL, and >10 ng/mL, concentrations below the lower limit of quantification were entered as 0 ng/mL.
Time Frame: 24 hours post dose on Week 6, Week 24, Week 48, Week 72, Week 96, Week 144, and Week 240
Population: The analysis was performed in the Safety Set population. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus (Core Period) | Everolimus (Extension Period)
Number analyzed (Participants) | 78 | 111
ng/mL
  Week 6 (n= 64, 94) | 5.8 (3.68) | 6.09 (3.708)
  Week 24 (n= 64, 89) | 6.59 (3.43) | 6.86 (3.504)
  Week 48 (n= 23, 86) | 7.28 (3.11) | 7.07 (3.214)
  Week 72 (n= 4, 92) | 6.08 (2.19) | 7.25 (3.66)
  Week 96 (n= 0, 83) | NA (NA) — No participant was evaluable, so value was not available. | 7.09 (3.697)
  Week 144 (n= 0, 69) | NA (NA) — No participant was evaluable, so value was not available. | 7.28 (3.35)
  Week 240 (n= 0, 13) | NA (NA) — No participant was evaluable, so value was not available. | 5.85 (2.507)

11. Secondary Outcome: Percentage of Participants With Renal Impairment During Core Period
Description: Renal function was assessed using glomerular filtration rate (GFR) based on age measure; Modification of Diet in Renal Disease (MDRD) formula for participants aged 18 years or older, defined as GFR equal to 32788*(serum creatinine (micromol/L)^-1.154)*(age^-0.203 )*(0.742, if female)*(1.210, if black), and Schwartz formula for participants less than 18 years defined as GFR equal to 0.41*height (cm)/ Serum creatinine (mg/dL). Participants with severe renal impairment defined as GFR < 30 mL/min/1.73 m^2 and participants with National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade 3/4 serum creatinine were reported.
Time Frame: Day 1 up to 28 days after end of treatment (Core period)
Population: The analysis was performed in the SAF population. Here, "Number of participants analysed" signifies the participants assessed for renal function during the study for each arm, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (Core Period) | Placebo (Core Period)
Number analyzed (Participants) | 78 | 39
Percentage of participants
  Grade 3 or 4 | 0 | 0
  Grade 1 or 2 | 3.8 | 0
  Grade 0 | 96.2 | 100

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were monitored from date of First Participant First Visit (FPFV) until Last Participant Last Visit (LPLV), 48 weeks and all other adverse events are monitored from First Participant First Treatment (FPFT) until LPLV, up to 4 years.
Description: For safety, the reporting arms have been created on the basis of actual exposure to study treatment
Groups:
- Everolimus Treated (Core and Extension Period): Participants who received everolimus treatment in core period and continued to receive evrolimus treatment in extension period.
- Placebo (Core) Then Everolimus Treated (Extension Period): Participants who received placebo in core period and then received evrolimus treatment in extension period.
- Placebo Treated (Core Period): Participants who received placebo in core period.
Arm/Group | Everolimus Treated (Core and Extension Period) | Placebo (Core) Then Everolimus Treated (Extension Period) | Placebo Treated (Core Period)
Serious Adverse Events (participants affected / at risk) | 33/78 | 17/33 | 3/6
Other Adverse Events (participants affected / at risk) | 77/78 | 33/33 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Treated (Core and Extension Period) (N=78) | Placebo (Core) Then Everolimus Treated (Extension Period) (N=33) | Placebo Treated (Core Period) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0
Ear infection bacterial (Infections and infestations) | 1 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 2 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pertussis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 11 | 5 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 4 | 1 | 2
Drooling (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 2 | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary pneumatocele (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Treated (Core and Extension Period) (N=78) | Placebo (Core) Then Everolimus Treated (Extension Period) (N=33) | Placebo Treated (Core Period) (N=6)
Anaemia (Blood and lymphatic system disorders) | 6 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 3 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 0
Constipation (Gastrointestinal disorders) | 11 | 2 | 0
Dental caries (Gastrointestinal disorders) | 5 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 7 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 33 | 6 | 0
Nausea (Gastrointestinal disorders) | 7 | 1 | 0
Oral pain (Gastrointestinal disorders) | 4 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 29 | 21 | 1
Toothache (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 24 | 6 | 1
Asthenia (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 16 | 2 | 0
Pyrexia (General disorders) | 25 | 7 | 2
Seasonal allergy (Immune system disorders) | 5 | 5 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 14 | 5 | 1
Cellulitis (Infections and infestations) | 4 | 0 | 0
Conjunctivitis (Infections and infestations) | 7 | 5 | 0
Croup infectious (Infections and infestations) | 4 | 0 | 0
Ear infection (Infections and infestations) | 14 | 4 | 0
Fungal infection (Infections and infestations) | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 4 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 9 | 4 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 2 | 0
Gastrointestinal viral infection (Infections and infestations) | 4 | 1 | 0
Influenza (Infections and infestations) | 6 | 2 | 0
Laryngitis (Infections and infestations) | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 30 | 15 | 1
Oral candidiasis (Infections and infestations) | 2 | 0 | 1
Otitis media (Infections and infestations) | 16 | 5 | 0
Pharyngitis (Infections and infestations) | 12 | 7 | 0
Pharyngitis streptococcal (Infections and infestations) | 15 | 2 | 1
Pneumonia (Infections and infestations) | 12 | 3 | 1
Respiratory tract infection (Infections and infestations) | 6 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 7 | 3 | 0
Rhinitis (Infections and infestations) | 8 | 2 | 0
Sinusitis (Infections and infestations) | 17 | 4 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 23 | 7 | 3
Urinary tract infection (Infections and infestations) | 7 | 1 | 0
Varicella (Infections and infestations) | 4 | 0 | 0
Viral infection (Infections and infestations) | 6 | 3 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 4 | 0
Excoriation (Injury, poisoning and procedural complications) | 4 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 4 | 1 | 0
Blood cholesterol increased (Investigations) | 11 | 3 | 1
Blood fibrinogen decreased (Investigations) | 5 | 6 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 6 | 0 | 0
Blood triglycerides increased (Investigations) | 7 | 0 | 0
Carbon dioxide decreased (Investigations) | 4 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 4 | 1 | 0
Low density lipoprotein increased (Investigations) | 6 | 2 | 1
Neutrophil count decreased (Investigations) | 6 | 1 | 0
Weight decreased (Investigations) | 5 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Convulsion (Nervous system disorders) | 31 | 13 | 4
Dizziness (Nervous system disorders) | 6 | 3 | 0
Epilepsy (Nervous system disorders) | 3 | 2 | 1
Headache (Nervous system disorders) | 13 | 6 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 6 | 0 | 0
Aggression (Psychiatric disorders) | 10 | 3 | 0
Agitation (Psychiatric disorders) | 6 | 1 | 0
Anxiety (Psychiatric disorders) | 10 | 3 | 0
Insomnia (Psychiatric disorders) | 11 | 4 | 0
Irritability (Psychiatric disorders) | 5 | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 5 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 3 | 0
Amenorrhoea (Reproductive system and breast disorders) | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 10 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 18 | 4 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 2 | 0
Hypertension (Vascular disorders) | 11 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.